CLINICAL TRIAL: NCT05273710
Title: Comparison of the Effects of Dietary Folate and Phytate on the Absorption of Zinc From Either Zinc-amino Acids (ZnAA) or Zinc-chloride (ZnCl2)
Brief Title: Effects of Dietary Folate and Phytate Zinc Absorption: Zinc Amino Acid Complexes vs. Zinc-chloride
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2020-01-12879
Record Dates: First submitted 2022-03-01; First posted 2022-03-10 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Dietary Zinc Absorption

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zinc absorption study (Other): Zinc absorption is determined from each of 3 test meals in all subjects.
  Interventions: Other: Regular toast and juice; Other: High phytate toast and juice; Other: Regular toast and juice, with folic acid

INTERVENTIONS:
Other: Regular toast and juice — Participants consume a single test meal composed of regular whole wheat toast and apple juice, and zinc absorption is measured.
Other: High phytate toast and juice — Participants consume a single test meal composed of high phytate whole wheat toast and apple juice, and zinc absorption is measured.
Other: Regular toast and juice, with folic acid — Participants consume a single test meal composed of regular whole wheat toast and apple juice, with 400 mcg folic acid; and zinc absorption is measured.

SUMMARY:
The purpose of this study is to determine the effects of consuming a small breakfast of juice and toast with added phytate or with taking a folic acid supplement on the absorption of a small amount of zinc that is either bound to amino acids or to chloride or picolinate. The results of this study will provide new information on how components of diet (e.g., phytate, and folic acid) affect the absorption of different forms of dietary zinc (e.g., zinc bound to amino acids, zinc chloride, and zinc picolinate).

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy men (i.e., have no current health issues requiring medications or a specific diet), 19 to 50 years of age, with a body mass index between 18 and 30 kg/m2, and willing to eat only the foods provided by the study for 17 days

Exclusion Criteria:

* Those reporting current chronic or acute diseases or HIV diagnosis, food allergies, smoking tobacco or marijuana, alcohol abuse, any contraindication to venipuncture such as bleeding disorders or use of blood thinners; use of illicit drugs; regular consumption of medications, micronutrient supplements, or both. Vegetarians, or those unable to eat meat, are also excluded since the foods for the study contain meat.

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2022-11-16 (Actual); Study Completion 2022-11-16 (Actual)

PRIMARY OUTCOMES:
Fractional zinc absorption | 48 hours
  Oral zinc tracer to tracee ratio in plasma, as a fraction of intravenous zinc tracer to tracee ratio

CONTACTS AND LOCATIONS:
Overall Officials: Janet C King, Ph.D., Principal Investigator — University of California, Berkeley
Locations (1):
- University of California, Berkeley, California, United States